CLINICAL TRIAL: NCT04463914
Title: Development and Testing of a Behavioral Activation Mobile Therapy for Elevated Depressive Symptoms
Brief Title: Evaluation of a Mobile Therapy for Elevated Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Dahne, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00096156; 5R42MH108219-04 (NIH)
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Depressive Symptoms; Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A- Treatment as Usual (Other): Participants in the treatment as usual group will be provided educational material about mood management available via the EHR with the suggestion to discuss questions with their PCP. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Interventions: Behavioral: Treatment as Usual
- Group B- Moodivate (Experimental): Participants randomized to the Moodivate condition will be instructed to utilize Moodivate regularly, at least once per day, for the treatment of depressed mood. Participants in the Moodivate group will receive a download code to download the Moodivate mobile application. Moodivate is a mobile app for individuals with elevated symptoms of depression. Within the app, users identify values, create activities, schedule activities, and rate mood daily. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Interventions: Behavioral: Behavioral Activation Therapy app
- Group C- Moodivate + EHR (Experimental): Participants randomized to the Moodivate + EHR condition will receive similar instructions as those randomized to Moodivate, but will also be instructed that their PCP will have access to metrics related to their app utilization and may choose to follow-up with them regarding treatment utilization and response. The PCP for each participant randomized to this condition will be provided EHR access to Moodivate metrics which will include metrics related to change in mood, frequency of app utilization, and frequency of activity completion. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Interventions: Behavioral: Behavioral Activation Therapy app + EHR

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy app — Moodivate focuses on tracking daily activities, recording daily mood, and identifying new activities to complete that may help improve mood. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Arms: Group B- Moodivate
Behavioral: Behavioral Activation Therapy app + EHR — Moodivate focuses on tracking daily activities, recording daily mood, and identifying new activities to complete that may help improve mood. The participant's primary care provider at MUSC will be provided access to a Moodivate provider portal that was developed by study team. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Arms: Group C- Moodivate + EHR
Behavioral: Treatment as Usual — Participants will be provided educational material about mood management available via the EHR with the suggestion to discuss questions with their PCP. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Arms: Group A- Treatment as Usual

SUMMARY:
The purpose of this research study is to evaluate a mobile application (app) for depression treatment. Participants will be randomly assigned to either receive the mobile app, "Moodivate", or not. If provided with Moodivate, participants will be asked to use the app regularly, at least once per day, throughout the study duration. Participants will be asked to complete electronic questionnaire measures throughout the study period. Participation in this study will take about 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Elevated depressive symptoms, defined as a score of > 10 on the Patient Health Questionnaire-9 (PHQ-9)57
* Age 18+
* Currently own an iOS- or Android-compatible smartphone
* Report willingness to utilize a mobile app for the treatment of depressed mood (response of "yes" on yes/no item)
* Have a current, valid e-mail address that is checked at least once per day or have regular access to text messages (to access follow-up assessments)
* Enrolled in Epic's MyChart program
* English fluency

Exclusion Criteria:

- Current suicidal ideation at study screening, defined as a response >1 (several days) on item nine of the PHQ-9 ("Over the last two weeks, how often have you been bothered by thoughts that you would be better off dead, or of hurting yourself?")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dahne, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahne J, Wahlquist AE, Carpenter MJ, Graboyes EM, Lejuez CW, Kustanowitz J, Natale N, Levins O, Player M, Diaz VA. A Digital Depression Treatment Program for Adults Treated in Primary Care: A Randomized Clinical Trial. JAMA Intern Med. 2025 Jun 1;185(6):692-701. doi: 10.1001/jamainternmed.2025.0494. PMID 40227715

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A- Treatment as Usual | Group B- Moodivate | Group C- Moodivate + EHR
Started | 212 | 216 | 221
Completed | 212 | 216 | 221
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A- Treatment as Usual | Group B- Moodivate | Group C- Moodivate + EHR | Total
Number analyzed (Participants) | 212 | 216 | 221 | 649
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.27 (15.83) | 44.53 (15.04) | 44.26 (14.84) | 44.68 (15.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 163 | 168 | 495
  Male | 48 | 53 | 53 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 16 | 40
  Not Hispanic or Latino | 200 | 204 | 205 | 609
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 3 | 3 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 51 | 47 | 39 | 137
  White | 148 | 153 | 169 | 470
  More than one race | 9 | 11 | 12 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Depressive Symptoms
Description: Patients will self report depressive symptoms weekly for 8 weeks with final follow-up at 12-weeks via the Beck Depression Inventory-II. The range of scores possible are 0 - 63, where lower scores are indicative of lower symptoms of depression.
Time Frame: Between baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A- Treatment as Usual | Group B- Moodivate | Group C- Moodivate + EHR
Number analyzed (Participants) | 212 | 216 | 221
score on a scale | -5.95 (11.61) | -11.24 (11.67) | -10.69 (12.87)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Group A- Treatment as Usual | Group B- Moodivate | Group C- Moodivate + EHR
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/216 | 0/221
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/216 | 0/221
Other Adverse Events (participants affected / at risk) | 0/212 | 0/216 | 0/221

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT04463914/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT04463914/ICF_000.pdf